CLINICAL TRIAL: NCT00427336
Title: Purine Analog-Based Conditioning for Allogeneic Stem Cell Transplantation in Patients With Severe Aplastic Anemia
Brief Title: Purine Analog-Based Conditioning in Patients With Severe Aplastic Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDP00-266
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2011-10-27 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-09

CONDITIONS: Aplastic Anemia
Keywords: Severe Aplastic Anemia; Bone Marrow Failure; Stem Cell Transplantation; Fludarabine; Cyclophosphamide; Antithymocyte Globulin; SAA; ATG; Cytoxan; Neosar; Fludarabine Phosphate; Thymoglobulin
MeSH Terms: conditions — Anemia, Aplastic; Bone Marrow Failure Disorders | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fludarabine + Cyclophosphamide + ATG (Experimental): Fludarabine 30 mg/m^2/day by vein (IV), Cyclophosphamide IV 300 mg/m^2/day, ATG (Antithymocyte Globulin) IV 3.75 mg/kg/day
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Antithymocyte Globulin

INTERVENTIONS:
Drug: Fludarabine — 30 mg/m^2 by vein daily over 30 minutes
  Other Names: Fludarabine Phosphate; Fludara
Drug: Cyclophosphamide — 300 mg/m^2 by vein daily over 2 hours
  Other Names: Cytoxan; Neosar
Drug: Antithymocyte Globulin — 3.75 mg/kg by vein daily over 4 hours
  Other Names: ATG; Thymoglobulin

SUMMARY:
Primary Objectives:

1. To determine the feasibility and toxicity of employing purine-analog based conditioning for allogeneic donor stem cell transplantation in patients with severe aplastic anemia (AA).
2. To determine the engraftment kinetics and degree of chimerism that can be achieved with this strategy.

DETAILED DESCRIPTION:
Before treatment starts, patients will have their bone marrow checked and will have lung, heart, and kidney tests.

Patients in this study will receive the drugs fludarabine, cyclophosphamide, and antithymocyte globulin by vein through a previously inserted plastic catheter that extends into the large chest vein. Fludarabine will be given daily for four days, cyclophosphamide will given daily for four days, and antithymocyte globulin will be given daily for four days (three days for related donor transplants).

Two days after the last dose of cyclophosphamide, donor marrow or stem cells will be infused through a catheter (thin plastic tube). Drugs will be given to lower the chance of an allergic reaction to the stem cells. Patients will also get shots of filgrastim (a drug that helps white blood cell growth) and antibiotics by mouth. The blood cell counts will fall to low levels during the first 2 weeks when patients may need transfusions of red blood cells and platelets. The chemotherapy will be given in the hospital. After the infusion of stem cells, patients will be monitored in the hospital. They will later be closely followed as outpatients and will be required to remain in the Houston area for about three months after the transplant.

Drugs (cyclosporine and methotrexate) to lower the chance of graft-versus-host disease will be given. Cyclosporine will be given as a continuous infusion starting 2 days before transplantation. Methotrexate will be given through the catheter on Days 1, 3, 6 and 11 after transplantation. Cyclosporine will be given as pills when the patient is able to swallow. Cyclosporine will be continued for no less than 6 months after transplantation after which it will be gradually stopped. The drug tacrolimus may be used instead of cyclosporine.

Blood, urine, bone marrow, and x-ray exams will be done as needed to monitor the results of bone marrow transplantation. Patients may require blood and platelet transfusions. Blood tests will be done daily while hospitalized and several times a week until the blood counts recover. Bone marrow aspiration and biopsies will be performed before the transplant, when the donated cells show signs of engraftment, and at other times during the next 1 to 3 years. They will be done to evaluate the growth of the transplant marrow, possible recurrence of malignancy, and recovery of immunity. If this treatment proves unsuccessful in more than three of the first ten patients, the study will be stopped.

This is an investigational study. The FDA has approved all of the drugs in this study for other indications. Up to 30 patients will be treated on this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients up to 70 years of age with a diagnosis of severe AA (Camitta et al., 1979) and a matched unrelated donor who are unresponsive to IS or who have relapsed after an initial response to IS. Patients with a diagnosis of SAA and an human leukocyte antigen (HLA) - compatible sibling donor are eligible only if they are 40 years of age or older (up to age 70) and regardless whether they have received IS or not. Patients with primary or secondary graft failure following autologous or allogeneic stem cell transplant are eligible.
* Patients must have a serum bilirubin of 2 mg/dl or less, serum creatinine < 2.0 mg/dl, no symptomatic cardiac or pulmonary disease and a PS of no more than 2. Life expectancy not severely limited by concomitant illness (> 12 weeks). Left ventricular ejection fraction > 40%, no uncontrolled arrhythmia or symptomatic cardiac disease. Forced Expiratory Volume in 1 Second (FEV1), Forced Vital Capacity (FVC) and Carbon Monoxide Diffusing Capacity (DLCO) > 40%. No symptomatic pulmonary disease. Negative pregnancy test.
* Patients must have an HLA-compatible related or unrelated donor willing to donate marrow or rhG-CSF-mobilized peripheral blood stem cells. In the event of transplants from matched unrelated donors, a high-resolution allele match for HLA-A, -B, -C, -DRB1 and DQB1 ("10 of 10 match") is preferred. However, a one-antigen mismatch ("micromismatch") is also considered acceptable matching ("9 of 10 match").
* Patients must sign informed consent. In the event of a pediatric patient (i.e., a minor), consent will be provided by their guardian/parent.
* Lack of clonal cytogenetic abnormalities associated with acute myeloid leukemia (AML), myelodysplastic syndrome (MDS) or other hematologic malignancies.

Exclusion Criteria:

* Life expectancy of less than 8 weeks. Inability to provide informed consent.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2000-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Anderlini, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 2000 to August 2009. All participants recruited at UT MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Fludarabine + Cyclophosphamide + ATG
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fludarabine + Cyclophosphamide + ATG
Number analyzed (Participants) | 9
Age Continuous [Median (Full Range); unit: years] | 39 [18 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Engraftment Response
Description: Engraftment defined as (1) the first of three consecutive days of an Absolute neutrophil count (ANC) >500/mL (b) the first of seven consecutive days of an unsupported platelet count 20,000. Patient needs to survive at least 28 days to be evaluable for engraftment. Chimerism studies need to demonstrate donor-derived hematopoiesis (>90%)
Time Frame: First 100 days post transplant.
Measure: Number; unit: Participants
Arm/Group | Fludarabine + Cyclophosphamide + ATG
Number analyzed (Participants) | 9
Participants | 9

ADVERSE EVENTS:
Time Frame: 7 years, 10 months
Arm/Group | Fludarabine + Cyclophosphamide + ATG
Serious Adverse Events (participants affected / at risk) | 6/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fludarabine + Cyclophosphamide + ATG (N=9)
Elevated Bilirubin (Hepatobiliary disorders) | 3 (3)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Elevated Creatinine (Renal and urinary disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Fever (Infections and infestations) | 1 (1)
Elevated Transaminases (Hepatobiliary disorders) | 1 (2)
Hypotension (Cardiac disorders) | 1 (1)
Headache (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fludarabine + Cyclophosphamide + ATG (N=9)
Nausea (Gastrointestinal disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Fever (Infections and infestations) | 2 (2)
Mucositis (Gastrointestinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Infection (Infections and infestations) | 1 (2)
Elevated Bilirubin (Hepatobiliary disorders) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Elevated Creatinine (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No